CLINICAL TRIAL: NCT02255929
Title: Gamma Knife Thalamotomy for Treatment of Essential Tremor
Brief Title: Gamma Knife Radiosurgery for Treatment of Essential Tremor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR 5585
Record Dates: First submitted 2014-09-17; First posted 2014-10-03 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Essential Tremor
Keywords: Benign Essential Tremor; Tremor; Neurologic Manifestations; Nervous System Diseases; Movement Disorders; Central Nervous System Diseases
MeSH Terms: conditions — Essential Tremor; Tremor; Neurologic Manifestations; Nervous System Diseases; Movement Disorders; Central Nervous System Diseases | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gamma Knife Radiosurgery (Experimental): Gamma Knife treatment is conducted in one day and takes approximately 70 to 90 minutes.
  Interventions: Radiation: Gamma Knife Radiosurgery

INTERVENTIONS:
Radiation: Gamma Knife Radiosurgery

SUMMARY:
The purpose of this study is to examine effects (good and bad) of gamma knife radiosurgery for essential tremor. The gamma knife places a small lesion in the brain to suppress tremors.

DETAILED DESCRIPTION:
This research is being done because although multiple studies evaluating gamma knife for essential tremor show good results, few studies evaluating patients prospectively have been done. Prior studies have looked at patient outcomes following treatment - also known as retrospective studies. In this study, data collection will initiate before treatment, to obtain consistent baseline evaluations from all study participants undergoing the gamma knife treatment and at specific intervals following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or older
* Diagnosis of essential tremor as confirmed from clinical history and examination by a neurologist or neurosurgeon
* Tremor following prior first line therapy with either propranolol or primidone
* Must be able to undergo MRI of brain and CT of head for treatment planning
* Postural or intention tremor severity score of greater than or equal to 2 in one hand/arm as measured by the CRST rating scale

Exclusion Criteria:

* Prior ipsilateral stereotactic radiosurgical ablation of the thalamus, ipsilateral deep brain stimulation, radiofrequency ablation of a ipsilateral thalamic target, or ultrasound ablation of an ipsilateral thalamic target
* Prior whole brain radiation therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Effectiveness based on Clinical Rating Scale for Tumor (CRST-Part B) questionnaires. | Baseline, 6, 12, 24, and 36 Months Post Treatment
  The change observed is represented by a writing and drawing score assessment of tremors. The assessment is conducted by a movement disorder neurologist in a blinded fashion.

SECONDARY OUTCOMES:
Safety Based on the Number of Incidences and Severity of Adverse Events Related with Gamma Knife Thalamotomy | Baseline, 6, 12, 24, and 36 Months Post Treatment
  Adverse Events to be reported as mild, moderate or severe

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Loiselle, MD, Principal Investigator — Swedish Medical Center Radiosurgery Center
Locations (1):
- Swedish Medical Center Radiosurgery Center, Seattle, Washington, United States

REFERENCES:
- See also: Click here for more information about the Swedish Medical Center Radiosurgery Center — http://www.swedish.org/services/radiosurgery-center